CLINICAL TRIAL: NCT04300322
Title: The Effectiveness of Cervical Pessary Versus Vaginal Progesterone for the Prevention of Preterm Birth in Women With Singleton Pregnancies and Short Cervix: a Multicenter Randomized Controlled Trial
Brief Title: Pessary Versus Progesterone in Singletons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: My Duc Phu Nhuan Hospital HCMC, Vietnam (Unknown); Quang Ninh Obstetrics and Pediatrics Hospital, Quang Ninh, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CS/BVMD/20/04
Record Dates: First submitted 2020-02-28; First posted 2020-03-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Preterm Birth; Short Cervix
Keywords: Preterm Birth; Singleton Pregnancies; Short Cervix; Pessary; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either pessary or progesterone in a 1:1 ratio with a variable block size of 2, 4 or 6.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical pessary (Active Comparator): Cervical pessary (Arabin) will be inserted to participants at 16-22 weeks and removed at 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Device: Cervical pessary
- Vaginal Progesterone (Active Comparator): Vaginal progesterone (Cyclogest 200 mg) once a day will be used, from 16-22 to 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Drug: Vaginal Progesterone

INTERVENTIONS:
Device: Cervical pessary — Arabin (cervical pessary) will be inserted at 16-22 weeks and removed at 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort
  Other Names: Arabin
  Arms: Cervical pessary
Drug: Vaginal Progesterone — Vaginal progesterone (Cyclogest 200 mg) once a day will be used, from 16-22 to 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Other Names: Cyclogest 200 mg
  Arms: Vaginal Progesterone

SUMMARY:
This study compares the effectiveness of cervical pessary to vaginal progesterone for prevention of preterm birth in women with singleton pregnancies and a cervix ≤25 mm.

Participants will be randomly assigned in a 1:1 ratio to receive cervical pessary or vaginal progesterone.

DETAILED DESCRIPTION:
This open label, multi-center, randomized controlled trial aims to compare the effectiveness of cervical pessary to vaginal progesterone for prevention of PTB in women with singleton pregnancies and a cervix ≤25 mm.

All women at 16 0/7 to 22 0/7 weeks with singleton pregnancies will undergo cervical length (CL) measurement and digital examination at screening routinely. Women with a CL ≤25 mm will be eligible for the study.

Subjects meeting the study criteria will be randomized into two groups: (1) treated with cervical pessary (Arabin) or (2) treated with 200 mg vaginal progesterone, once daily.

After written informed consent, women will be randomly assigned in a 1:1 ratio to receive a cervical pessary or progesterone. Assignment to treatment allocation will be done via a web portal hosted by HOPE Research Center, Vietnam. The randomization schedule will be computer-generated at HOPE Research Center, with a permuted random block size of 2, 4 or 6. Blinding will not be possible due to the nature of interventions.

For those who randomised to pessary group, a pessary certified by European Conformity (Arabin®, Dr Arabin GmbH & Co KG, Germany) will be inserted through the vagina, upward around the cervix by 2-4 senior clinicians, who had experienced with pessary used at each site, within one week of randomization.

Women allocated to progesterone group will be receiving 200 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 200 mg, Actavis, United Kingdom), once daily at bedtime. They will be given a monitoring sheet and instructed to note everyday the date of using.

In case of premature rupture of membranes, active vaginal bleeding, other signs of preterm labor or severe patient discomfort, the pessary may be removed. If participants develop (threatened) preterm labor, they will receive treatment per local protocol. Intervention will be stopped at 370/7 weeks of gestation or at delivery.

Along side with this trial, another study will be conducted to determine how changes in peripheral blood and cervical inflammatory markers are impacted by progesterone versus pessary. Because of that, participants will be asked to take 5 ml blood sample and cervical-vaginal discharge sampling at the time of randomization, 4-8 weeks after randomization and before giving birth.

A cost-effectiveness analysis will also be conducted alongside this RCT. Data will be reported in a separated paper.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Cervical length ≤ 25 mm, measured by TVS at the second-trimester ultrasonography (16 0/7-22 0/7 weeks of gestation)
* Not participating in any other study which has intervention on maternity or fetus at the same time
* Provision of written informed consent to participate as shown by a signature on the patient consent form.

Exclusion Criteria:

* Cervical dilation with visible amniotic membranes or amniotic membranes prolapsed into the vagina
* Major congenital abnormalities of the fetus
* Presence of severe vaginal discharge
* Presence of vaginitis or cervicitis
* Presence of vaginal bleeding
* Preterm premature rupture of membranes
* Premature labor without ruptured membrane at the time of screening
* Suspected chorioamnionitis
* Unable to have cervical pessary inserted
* Cerclage or pessary in place

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of preterm birth <37 weeks of gestation by any cause | From date of randomisation until 36 6/7 weeks
  Birth before 37 weeks

SECONDARY OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery
Time from randomization to delivery | From date of randomisation until the date of delivery.
  Time interval between randomisation and delivery
Rate of preterm birth before 28 weeks of gestation | From date of randomisation until 27 6/7 weeks
  Birth before 28 weeks
Rate of preterm birth before 34 weeks of gestation | From date of randomisation until 33 6/7 weeks
  Birth before 34 weeks
Rate of spontaneous preterm birth <28 weeks | From date of randomisation until 27 6/7 weeks
  Birth spontaneously before 28 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Rate of spontaneous preterm birth <34 weeks | From date of randomisation until 33 6/7 weeks
  Birth spontaneously before 34 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Rate of spontaneous preterm birth <37 weeks | From date of randomisation until 36 6/7 weeks
  Birth spontaneously before 37 weeks' gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Rate of iatrogenic preterm birth <28 weeks | From date of randomisation until 27 6/7 weeks
  Birth non-spontaneously before 28 weeks' gestation
Rate of iatrogenic preterm birth <34 weeks | From date of randomisation until 33 6/7 weeks
  Birth non-spontaneously before 34 weeks' gestation
Rate of iatrogenic preterm birth <37 weeks | From date of randomisation until 36 6/7 weeks
  Birth non-spontaneously before 37 weeks' gestation
Rate of onset of labor | At birth
  Spontaneous, labor induction, elective C-section
Rate of modes of delivery | At birth
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Rate of all live births at any gestational age | At birth
  The birth of at least one newborn, regardless of gestational age, that exhibits any sign of life such as respiration, heartbeat, umbilical pulsation or movement of voluntary muscles
Rate of use of tocolytic drugs | From 24 0/7 to 36 6/7 weeks' gestation
  Use of any tocolytic drug to treat preterm labour
Rate of use of antenatal corticosteroids | From 24 0/7 to 36 6/7 weeks' gestation
  Use of antenatal corticosteroids to prevent respiratory distressed syndrome
Rate of use of MgSO4 for neuroprotection | From 28 0/7 to 31 6/7 weeks' gestation
  Use of MgSO4 for neuroprotection
Rate of preterm premature rupture of membranes | From randomization to less than 37 weeks, up to 21 weeks
  Prelabour rupture of membranes and gestational age less than 37 weeks
Length of maternal admission for preterm labor (days) | From randomization to 37 week
  Number of admission days for treatment of preterm labour
Rate of chorioamnionitis | From randomization to delivery, up to 28 weeks
  Intraamniotic infection
Rate of maternal mortality | From randomization to delivery, up to 28 weeks
  Death of the mother
Birthweight (mean) | At birth
  Weight of baby born
Birthweight <1500 g | At birth
  Weight of baby born <1500g
Birthweight <2500 g | At birth
  Weight of baby born <2500g
Rate of congenital anomalies | At birth
  Any congenital anomalies detected in baby born
5-min Apgar score | At birth
  Apgar score at 5 minute after birth. 5-minute Apgar score of 7-10 as reassuring, a score of 4-6 as moderately abnormal, and a score of 0-3 as low in the term infant and late-preterm infant.
5-min Apgar score <7 | At birth
  Apgar score at 5 minute after birth <7. An increased relative risk of cerebral palsy.
Rate of admission to neonatal intensive care unit (NICU) | Up to 28 days of life after the due day
  Admission to neonatal intensive care unit of baby
Length of NICU admission | Up to 28 days of life after the due day
  Number of admission days to NICU
Rate of death before discharge | Up to 28 days of life after the due day
  Death of newborn before discharge from nursery
Rate of neonatal death | Up to 28 days of life after the due day
  Death of a live-born infant within the first 28 days of life after the due day
Rate of perinatal death | After 20 weeks of gestation to 28 days of life after the due day
  Intrauterine fetal death after 20 weeks of gestation, or neonatal death
Rate of stillbirth | After 20 weeks of gestation until the date of delivery
  Baby born with no signs of life at or after 20 weeks' gestation
Rate of composite of poor perinatal outcomes | Up to 28 days of life after the due day
  Foetal or neonatal death, intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis
Rate of respiratory distress syndrome | Up to 28 days of life after the due day
  presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Rate of periventricular haemorrhage II B or worse | Up to 28 days of life after the due day
  Repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al
Rate of necrotizing enterocolitis | Up to 28 days of life after the due day
  Diagnosed according to Bell
Rate of proven sepsis | Up to 28 days of life after the due day
  The combination of clinical signs and positive blood cultures
Rate of maternal vaginal side effects | From date of randomisation until delivery, which is up to 24 weeks
  Including vaginal discharge, vaginal bleeding, vaginal infection (confirmed by vaginal discharge culture)
Vaginal pain Score | From date of randomisation until delivery, which is up to 24 weeks
  Evaluated by VAS numerical rating scale. Assessments with units on a Scale.
Rate of pessary repositioning | From date of randomisation until delivery, which is up to 24 weeks
  After pessary initial placement, requiring to reposition the pessary by any reasons
Rate of maternal cervical side effects | From date of randomisation until delivery, which is up to 24 weeks
  Including necrosis or rupture of the cervix, cervical laceration

CONTACTS AND LOCATIONS:
Overall Officials: Vinh Q Dang, MD, Principal Investigator — Mỹ Đức Hospital
Locations (3):
- Vietnam (3):
  - My Duc Phu Nhuan Hospital, Ho Chi Minh City, Phu Nhuan
  - Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh
  - Quang Ninh Obstetrics and Pediatrics Hospital, Quang Ninh

REFERENCES:
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Platt MJ. Outcomes in preterm infants. Public Health. 2014 May;128(5):399-403. doi: 10.1016/j.puhe.2014.03.010. Epub 2014 May 1. PMID 24794180
- [Background] Lawn JE, Kinney MV, Belizan JM, Mason EM, McDougall L, Larson J, Lackritz E, Friberg IK, Howson CP; Born Too Soon Preterm Birth Action Group. Born too soon: accelerating actions for prevention and care of 15 million newborns born too soon. Reprod Health. 2013;10 Suppl 1(Suppl 1):S6. doi: 10.1186/1742-4755-10-S1-S6. Epub 2013 Nov 15. PMID 24625252
- [Background] Vogel JP, Chawanpaiboon S, Moller AB, Watananirun K, Bonet M, Lumbiganon P. The global epidemiology of preterm birth. Best Pract Res Clin Obstet Gynaecol. 2018 Oct;52:3-12. doi: 10.1016/j.bpobgyn.2018.04.003. Epub 2018 Apr 26. PMID 29779863
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; McIntosh J, Feltovich H, Berghella V, Manuck T. The role of routine cervical length screening in selected high- and low-risk women for preterm birth prevention. Am J Obstet Gynecol. 2016 Sep;215(3):B2-7. doi: 10.1016/j.ajog.2016.04.027. Epub 2016 Apr 28. PMID 27133011
- [Background] Leung TN, Pang MW, Leung TY, Poon CF, Wong SM, Lau TK. Cervical length at 18-22 weeks of gestation for prediction of spontaneous preterm delivery in Hong Kong Chinese women. Ultrasound Obstet Gynecol. 2005 Dec;26(7):713-7. doi: 10.1002/uog.2617. PMID 16308894
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Norman JE, Marlow N, Messow CM, Shennan A, Bennett PR, Thornton S, Robson SC, McConnachie A, Petrou S, Sebire NJ, Lavender T, Whyte S, Norrie J; OPPTIMUM study group. Vaginal progesterone prophylaxis for preterm birth (the OPPTIMUM study): a multicentre, randomised, double-blind trial. Lancet. 2016 May 21;387(10033):2106-2116. doi: 10.1016/S0140-6736(16)00350-0. Epub 2016 Feb 24. PMID 26921136
- [Background] Romero R, Conde-Agudelo A, Da Fonseca E, O'Brien JM, Cetingoz E, Creasy GW, Hassan SS, Nicolaides KH. Vaginal progesterone for preventing preterm birth and adverse perinatal outcomes in singleton gestations with a short cervix: a meta-analysis of individual patient data. Am J Obstet Gynecol. 2018 Feb;218(2):161-180. doi: 10.1016/j.ajog.2017.11.576. Epub 2017 Nov 17. PMID 29157866
- [Background] Arabin B, Halbesma JR, Vork F, Hubener M, van Eyck J. Is treatment with vaginal pessaries an option in patients with a sonographically detected short cervix? J Perinat Med. 2003;31(2):122-33. doi: 10.1515/JPM.2003.017. PMID 12747228
- [Background] Goya M, de la Calle M, Pratcorona L, Merced C, Rodo C, Munoz B, Juan M, Serrano A, Llurba E, Higueras T, Carreras E, Cabero L; PECEP-Twins Trial Group. Cervical pessary to prevent preterm birth in women with twin gestation and sonographic short cervix: a multicenter randomized controlled trial (PECEP-Twins). Am J Obstet Gynecol. 2016 Feb;214(2):145-152. doi: 10.1016/j.ajog.2015.11.012. Epub 2015 Nov 25. PMID 26627728
- [Background] Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, Brons J, Duvekot H, Bijvank BN, Franssen M, Gaugler I, de Graaf I, Oudijk M, Papatsonis D, Pernet P, Porath M, Scheepers L, Sikkema M, Sporken J, Visser H, van Wijngaarden W, Woiski M, van Pampus M, Mol BW, Bekedam D. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicentre, open-label randomised controlled trial. Lancet. 2013 Oct 19;382(9901):1341-9. doi: 10.1016/S0140-6736(13)61408-7. Epub 2013 Aug 5. PMID 23924878
- [Background] Dang VQ, Nguyen LK, Pham TD, He YTN, Vu KN, Phan MTN, Le TQ, Le CH, Vuong LN, Mol BW. Pessary Compared With Vaginal Progesterone for the Prevention of Preterm Birth in Women With Twin Pregnancies and Cervical Length Less Than 38 mm: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):459-467. doi: 10.1097/AOG.0000000000003136. PMID 30741812
- [Background] Jin Z, Chen L, Qiao D, Tiwari A, Jaunky CD, Sun B, Wang L, Yu H. Cervical pessary for preventing preterm birth: a meta-analysis. J Matern Fetal Neonatal Med. 2019 Apr;32(7):1148-1154. doi: 10.1080/14767058.2017.1401998. Epub 2017 Nov 20. PMID 29103351
- [Background] Saccone G, Ciardulli A, Xodo S, Dugoff L, Ludmir J, Pagani G, Visentin S, Gizzo S, Volpe N, Maruotti GM, Rizzo G, Martinelli P, Berghella V. Cervical Pessary for Preventing Preterm Birth in Singleton Pregnancies With Short Cervical Length: A Systematic Review and Meta-analysis. J Ultrasound Med. 2017 Aug;36(8):1535-1543. doi: 10.7863/ultra.16.08054. Epub 2017 Apr 11. PMID 28398701